CLINICAL TRIAL: NCT05004363
Title: Lokelma for Maximisation of RAAS Inhibition in CKD Patients With Heart Failure; Randomised.
Brief Title: Lokelma for RAAS Maximisation in CKD & Heart Failure.
Acronym: LIFT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St George's, University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020.0071; 2020-002946-18 (EudraCT Number)
Record Dates: First submitted 2020-06-08; First posted 2021-08-13 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Chronic Kidney Diseases; Heart Failure With Reduced Ejection Fraction; Hyperkalemia; ACE Inhibitor Induced Hyperkalaemia; Mineralocorticoid Resistant Hyperkalemia
Keywords: Acute Kidney Injury; Sodium Zirconium Cyclosilicate
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperkalemia; Pseudohypoaldosteronism; Acute Kidney Injury

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lokelma (Active Comparator): Lokelma therapy
  Interventions: Drug: Lokelma Oral Product
- Control (Placebo Comparator): Placebo
  Interventions: Drug: Lokelma Oral Product

INTERVENTIONS:
Drug: Lokelma Oral Product — Potassium binder
  Other Names: placebo

SUMMARY:
Background: CKD in patients with heart failure (HF) is common and associated with poor prognosis. Despite evidence of benefit with Renin-Angiotensin-Aldosterone-System inhibitor (RAASi) agents, they are avoided due to fear of hyperkalaemia. New potassium binders, e.g. Sodium Zirconium Cyclosilicate (SZC), reduce incidence of hyperkalaemia in CKD-HF patients and hence may help RAASi maximisation, which has not been investigated in an RCT.

Purpose: The proposed study will randomise HFrEF patients with stable CKD 3-5 and serum potassium 5-5.0 mmol/L, to receive SZC or placebo while RAASi therapy is maximised. The aim of the study is to examine if SZC is superior to placebo in achieving maximal doses of ACEi/ARB, e.g. Ramipril 10 mg, Candesartan 32 mg; and mineralocorticoid receptor antagonist, e.g. Epleronone 50 mg or Spironolactone 50 mg, avoiding hyperkalaemia.

Methods: Eligible patients with eGFR<60 mL/min/1.73m2, heart failure (EF<40%) on none/submaximal dose of RAASi will be randomised to receive 10g TDS of investigational medicinal product (IMP), either SZC or placebo, for 48 hours and in 10 or 5g OD guided by laboratory serum potassium (K+). Every two weeks the RAASi dose will be increased and IMP adjusted according to a strict protocol and guided by laboratory potassium and creatinine. The primary endpoint of the study is achievement of maximal dose of RAASi in randomised patients avoiding hyperkalaemia, i.e. K+≤5.6 mmol/L. Patients will be allowed to continue with RAASi maximisation to K+<6.0mmol/L. Patients will be tested at baseline and follow-up visits for hyperkalaemia, AKI, symptomatic hypotension and QT prolongation on ECG.

Results: The study results will show if SZC is superior to placebo for RAASi maximisation in CKD-HF patients while maintaining safe levels of serum potassium without any adverse impact on quality of life. The study will demonstrate if SZC allows higher RAASi dose and more dose escalations than placebo. It will also examine the impact of RAASi escalation on creatinine, proteinuria, and cardiac blood biomarkers.

Conclusion: If positive, the results of this study will demonstrate that SZC enables RAASi up titration in CKD-HF patients, which potentially can help achieve optimal treatment and improve quality of life of the patient.

DETAILED DESCRIPTION:
Title Lokelma for maximisation of RAAS inhibition in CKD patients with Heart Failure; RCT (LiFT) Clinical Phase Phase III Trial Design Double-Blind, Placebo-Controlled, Randomised Trial Participant Population Patients with systolic heart failure chronic kidney disease 3-5 and no/submaximal RAASi

Inclusion.Criteria: :

* Age >18 years
* Heart failure, clinical or echo confirmed (HFrEF); patients with AF will be included provided the EF can be determined
* NYHA class II to IV
* Serum potassium 5.0-5.5 mmol/L
* Adequate blood pressure (>90 mm Hg systolic and without postural hypotension; drop of Systolic Blood Pressure >20 or feeling dizzy with change in posture; exclude patients with symptomatic hypotension due to high doses of ACEi/ARB or MRA unless the clinical condition has improved)
* CKD with stable eGFR <60 ml/min/1.73m2
* None or submaximal dose of ACEi/ARB and/or MRA or both

Exclusion:

* Pregnancy
* Active malignancy or infection
* BMI>35 kg/m2
* Poorly controlled sugar HBA1C> 70 mmol/mmol
* Recent ACS
* Potassium therapy
* Prolonged QT>550msec, congenital QT syndrome and history of prolong QT requiring drug discontinuation Planned Sample Size/Target 130 patients

Treatment duration 2 to 12 weeks Follow up duration 4-14 weeks Planned Trial Period 18 months Objectives

Outcome Measures: see below for the primary and secondary outcomes, briefly the study aims compare Sodium Zirconium Cyclosilicate (SZC) and Placebo with respect to enabling patients to achieve the target Renin-Angiotensin-Aldosterone-System-inhibitors (RAASi) dose while keeping K+ < 5.6. (numbers and proportion of patients in each group)

Investigational Medicinal Product Sodium Zirconium Cyclosilicate

Formulation, Dose, Route of Administration Powdered, to be taken orally dissolved in water, 10 g TDS for 48 hours followed by 10 or 5 g per day

BACKGROUND Chronic Kidney disease (CKD) is common in patients with heart failure, 32% in a meta-analysis of 1,076,104 patients and 47% in all acute heart failure admissions in our hospital. [Damman,K. 2014] These patients suffer 2.4 times higher mortality. Potentially lifesaving medications for systolic heart failure are not used in patients with CKD and heart failure due to risk of hyperkalaemia. These medications include Angiotensin Converting Enzyme inhibitors (ACEi) or angiotensin receptor blockers (ARB) and mineralocorticoid receptor antagonists (MRA) [Bowling 2013; Eschalier,R. 2013]. The risk of hyperkalaemia in CKD stage 4-5 patients on ACEi and MRA is high and potentially fatal. [Sarafidis,P.A. 2012] Hence there is reluctance amongst general practitioners, general physicians and cardiologists managing these patients to use medications which may increase serum potassium [Epstein,M. 2015].

St George's experience:

In a study of 1056 acute heart failure admissions of 851 patients at St George's Hospital patients with CKD stage 4/5 and systolic heart failure were less likely to receive ACEi/ARB compared to no-CKD patients (36% versus 84%; p<0.001) and less likely to receive MRA (17% versus 57%; p<0.001) http://onlinelibrary.wiley.com/doi/10.1002/ehf2.12185/full [Jenkins,R. 2017]. These findings have led to the setting up of a kidney failure-heart failure service at St George's Hospital funded by three local clinical commissioning groups to improve care for these patients.

St George's Hospital has an established heart failure unit and more recently a kidney failure-heart failure service. Audit of all new referrals to our kidney failure-heart failure clinic between March and September 2017 have shown that only 3% of all patients with left ventricular systolic dysfunction was on maximum dose of ACEi/ARB, and only 2% was on maximum dose of MRA. In another audit of 200 patients with CKD followed in our heart failure clinics between 1 March and 5 October 2017 only 13% of patients were on maximum dose of ACEi/ARB and 2% on maximum dose of MRA.

Sodium Zirconium Cyclosilicate (SZC) for hyperkalaemia:

Recent studies have shown that Sodium Zirconium Cyclosilicate lowers serum potassium non-CKD, CKD and separately in heart failure patients [Ash,S.R. 2015; Packham,D.K. 2015; Kosiborod,M. 2014; Anker,S.D. 2015]. Another potassium binder has also been shown to be effective. In a phase 3 randomised controlled trial of 258 patients, Sodium Zirconium Cyclosilicate lowered serum potassium from 5.6 to 4.5 mmol/L in 48 hours and maintained a potassium of <5.1 mmol/L in 90% (as opposed to 48% of patients on placebo. Most potassium binder studies have been short and none have investigated exclusively the high-risk group with CKD and heart failure, particularly with an aim to maximise RAASi therapy.

Statistical outcome measure:

Achieving target level of RAASi without hyperkalaemia i.e. serum potassium of >5.6 mmol/L (and potassium>6.0 mmol//L)

Event definition:

The binary outcome is defined as reaching potassium level of >5.6 mmol/L within the trial period. Serum potassium will be measured by point of care and laboratory testing. For the extended study the event will be defined as a potassium>6.0 mmol/L.

TRIAL DESIGN We propose a pilot 1:1 randomised placebo-controlled clinical trial to investigate the effect of the potential drug aiming at lowering the potassium levels if taken in conjunction with RAASi. Randomisation is stratified by the baseline RAASi dose the patients are subjected to when they join the trial. All eligible patients will be randomised to either oral Lokelma or equivalent placebo.

The trial will consist of the following phases: screening, correction phase and maintenance phase. During screening, a patient's eligibility will be assessed. After the screening is completed, the eligible patients will be randomized to Lokelma or Placebo and the initial potassium correction phase will be initiated. This phase will use correction phase dosing as per label (10 mg thrice daily) and be at most 48h long. During this period, potassium will be assessed at 48 hours, and patients judged to be normokalaemic (K+ between 3.5 and 5) will be transferred to the maintenance phase and initiate maintenance phase dosing regimen. After 48h, all patients will be transferred to maintenance phase, regardless of whether or not they are found to be normokalaemic at that time point. During the maintenance phase, a titration of IP will take place as shown below.

In parallel to the IP administration, a patient's ACEi/ARB and MRA treatment will be initiated or, if a patient already on ACEi/ARB and MRA, intensified. For details, see Study Schema and below.

Consent Full informed consent will be obtained prior to the participant undergoing any activities that are specifically for the purposes of the study.

The participant's GP will be informed in writing of their participation in the study.

Baseline data Baseline data will be recorded on the eCRF (web based secure system "redcap") and will include demographics such as age, gender, ethnicity; clinical comorbidities such as diabetes, hypertension, ischaemic heart disease; cardiovascular risk factors such as hypercholesterolemia, BMI, smoking, family history of IHD; blood test results such as haemoglobin, ferritin, urea, creatinine, sodium, potassium, BNP, troponin, calcium, phosphate, PTH, ECG and results of an echocardiogram. In addition, we will record pulse, BP (average of 3), weight, oedema, chest crepitations, elevated Jugular Venous Pressure (JVP), frailty score, QOL score.

Trial assessments Patients will be seen every two weeks for safety checks, blood tests, drug dosing and RAASi dosing. Data will be recorded on history for symptoms of heart failure, breathlessness, tiredness, leg swelling; physical examination finding, weight, oedema, chest crackles; blood test sodium, potassium, creatinine and drug dose.

The end of trial visit will record the same along with the QOL score. Long term follow-up assessments At the end of the trial the patient's data will be collected from the EPR on RAASi dose and outcome from their standard of care visits. There will be no follow up visits related to the trial.

Withdrawal criteria The patient may be withdrawn from the study if they request to do so, or due to safety concerns (such as a SUSAR). Each withdrawal will be replaced. Their data will be collected from EPR until the end of the study. The study may need to be stopped if there are multiple SUSARs; this will be discussed with the DMC.

Storage and analysis of clinical (biological) samples The sample will be collected and serum/plasma will be saved in -80 degrees Celsius freezer in the cardiovascular research institute for future biochemical analysis.

End of trial The trial will end with the last visit for the last patient. The MHRA and the REC will be notified within 90 days of the trial end.

TRIAL TREATMENTS Lokelma or matching Placebo will be administered 10 g thrice daily for the initial 48h. If normokalaemia, defined as K+ between 3.5 and 5, is reached earlier, maintenance phase dosing will be initiated, starting with 5 g daily. If by the end of the correction phase normokalaemia is not reached, the patient will be started on 10 g daily dosing.

During the maintenance phase, the IP will be titrated as follows:

Dose at start of visit Serum potassium end of visit Dose change at the end of visit If on 10 g daily 5.0-6.0 mmol/l Continue 10 g daily 3.5-5.0 mmol/l Change to 5 g daily <3.5 mmol/l Stop >6 mmol/l Stop and initiate rescue If on 5 g daily >5.0 mmol/l Change to 10 g daily 3.5-5.0 mmol/l Continue 5 g daily <3.5 mmol/l Stop If on 0 g daily (temporary stop) <= 5 Continue with no IP >5 Initiate 5 g daily

The drug can be restarted 2 weeks after discontinuation due to hypokalaemia depending on the blood result.

A patient will remain on their baseline RAASi treatment during the first two weeks post-randomization. The dose of RAASi will then be increased in a step-wise fashion as mentioned above every two weeks provided there is no allergy, severe hyperkalaemia (potassium >6.0 mmol/L) or symptomatic hypotension.

In case of allergy or severe hyperkalaemia are observed, the RAASi treatment will be stopped with no possibility of re-initiation. In case of symptomatic hypotension, the change in dosing will be delayed. The dose changes will be allowed within 2 days of the scheduled visit.

Other concomitant treatments and monitoring Other concomitant medications will continue. During the trial period clinicians are advised to use diuretics such as furosemide for lung congestion, shortness of breath and oedema in doses 40-160 mg daily (or equivalent bumetanide 1-4 mg), and metolazone 2.5 to 5 mg daily as clinically indicated. Patients will be encouraged to monitor their own blood pressures at home.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Heart failure, clinical or echo confirmed (HFrEF); patients with AF will be included provided the EF can be determined
* NYHA class II to IV
* Serum potassium 5.0-5.5 mmol/L
* Adequate blood pressure (>90 mm Hg systolic and without postural hypotension; drop of Systolic Blood Pressure >20 or feeling dizzy with change in posture; exclude patients with symptomatic hypotension due to high doses of ACEi/ARB or MRA unless the clinical condition has improved)
* CKD with stable eGFR <60 ml/min/1.73m2
* None or submaximal dose of ACEi/ARB and/or MRA or both

Exclusion Criteria:

* • Pregnancy

  * Active malignancy or infection
  * BMI>35 kg/m2
  * Poorly controlled sugar HBA1C> 70 mmol/mmol
  * Recent ACS
  * Potassium therapy
  * Prolonged QT>550msec, congenital QT syndrome and history of prolong QT requiring drug discontinuation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2022-01-19 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants who achieve the maximum dose | 16 weeks
  Ramipril 5 mg OD + Spironolactone 25 mg OD for patients on a baseline RAASi dose that is less than Ramipril 5 mg OD + Spironolactone 25 mg OD or equivalent Ramipril 10 mg OD + Spironolactone 50 mg OD for patients on a baseline RAASi dose that is more or equal than Ramipril 5 mg OD + Spironolactone 25 mg OD or equivalent

SECONDARY OUTCOMES:
Number of participants achieving other outcomes | 16 weeks
  1. Achieving maximum dose of Mineralocorticoid receptor antagonists (MRA) and Angiotension-converting enzyme (ACEi) / Angiotensin-receptor blockers (ARB) and K+<5.6 mmol/L
  2. Achieving maximum dose of MRA and ACEi/ARB and K+≤6.0 mmol/L
  3. Time since randomisation to first occurrence of hyperkalaemia (K+>5.5 mmol/L)
  4. Time since randomisation to severe hyperkalaemia (K+>6.0)
  5. Number of ACEi/ARB, MRA end of study as compared to baseline
  6. Number of hospital admissions and duration of hospital admissions during the study
  7. Change in serum potassium at the respective visits as compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Debasish Banerjee, MD FRCP, Principal Investigator — St Georges's, University of London
Locations (1):
- St Georges, University of London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
It will be shared by study team, TSC, DSMB